CLINICAL TRIAL: NCT02024334
Title: Study of Therapeutic Effects and Side Effects of Leflunomide in Methotrexate Refractory Juvenile Idiopathic Arthritis
Brief Title: Efficacy Study of Leflunomide to Treat Juvenile Idiopathic Arthritis
Acronym: JIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rezaieyazdi, Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 900527
Record Dates: First submitted 2013-12-10; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA; LEFLUNOMIDE; EFFICACY
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Leflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- leflunomide (Active Comparator): leflunomide tablet: for patients less than 20 kg: 10 mg every 2 day, for patients 20 - 40 kg: 10 mg daily, for patients more than 40 kg: 20 mg daily.
  Interventions: Drug: Leflunomide
- placebo (Placebo Comparator): placebo tablet for patients less than 20 kg: 10 mg every 2 day, for patients 20 - 40 kg: 10 mg daily, for patients more than 40 kg: 20 mg daily.

INTERVENTIONS:
Drug: Leflunomide
  Other Names: arava
  Arms: leflunomide

SUMMARY:
A randomized double blind clinical trial to assess efficacy of leflunomide in treatment of refractory juvenile idiopathic arthritis.

Patients are randomly divided into two groups. In group 1 leflunomide and in group 2 placebos will be added to conventional treatment for three months. therapeutic responses will be evaluated by ACRpedi (American College of Rheumatology Pediatric) scores every 4 weeks.

DETAILED DESCRIPTION:
30 Patients(2-19 y) are randomly divided into two groups. In group 1 leflunomide will be added to conventional treatment, 5-20 mg daily based on weight.

In group 2 placebo will be prescribed as same as leflunomide. The course of treatment is 3 months. Every 4 weeks ACRped 30, 50, 70 should be determined to evaluate therapeutic response. Side effects of treatment will be assessed by physical examination and lab tests every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* JIA based on ACR criteria
* age between 2- 19 y
* polyarticular, oligoarticular(> or = 3 active joints) or extended oligoarticular subtypes
* resistance to conventional treatment

Exclusion Criteria:

* pregnancy
* malignancy
* severe active infection
* other rheumatic diseases or overlap
* ALT(Alanine transaminase) or bilirubin > 3 folds
* IVIG (Intravenous immunoglobulin) treatment during last 2 weeks
* biologic agents during last 3 months

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
thirty percent changes in the ACR Pediatric core set of disease activity measures in at least three of the six response variables (ACR Pedi 30) | baseline, week 4, week 8, week 12
  6 variables including: number of joints with arthritis, number of joints with limited range of motion, physician assessment, patient assessment, ESR (Erythrocyte Sedimentation Rate), CHAQ (Childhood Health Assessment Questionnaire) score.

SECONDARY OUTCOMES:
50% and 70% changes in the ACR Pediatric core set of disease activity measures in at least three of the six response variables (ACR Pedi 30) | baseline, week 4, week 8, week 12
  6 variables including: number of joints with arthritis, number of joints with limited range of motion, physician assessment, patient assessment, ESR, CHAQ score.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Rezaieyazdi, MD, Principal Investigator — Rheumatic Diseases Research Center, Ghaem Hospital, School of Medicine, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Mashhad, Khorasan Razavi, Iran